CLINICAL TRIAL: NCT03531489
Title: Pilot, Single Center Study of Ambulatory Respiratory Assist Device in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Study of Ambulatory Respiratory Assist Device in Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Right-Air (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Penn 826372
Record Dates: First submitted 2018-04-16; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Part 1: Feasibility (Experimental): Patients will perform 6-minute walk test with AIR-AD to allow for observation and real-time feedback.
  Interventions: Device: AIR-AD
- Part 2: Crossover (Experimental): Crossover design where investigator will compare wearing of AIR-AD during exercise to compare distance walked with and without it.
  Interventions: Device: AIR-AD

INTERVENTIONS:
Device: AIR-AD — Non-significant risk medical device as decided by institutional review board

SUMMARY:
The study is a two-part small scale, open-label, pilot study to evaluate feasibility and proof-of-concept for a respiratory assist medical device. The study population will consist of severe Chronic Obstructive Pulmonary Disease (COPD) subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe COPD (by ATS criteria)

1. FEV1/FVC <0.70
2. FEV1 < 60% Predicted

Exclusion Criteria:

1. Physical limitation that prevents walking for 6 minutes (e.g. lower extremity amputation, arthritis limiting function, significant angina, etc…)
2. Lung pathology not explained by COPD, which may limit functional capacity (e.g. pulmonary fibrosis, malignancy, history of lung reduction surgery, etc…)
3. Pregnancy
4. Age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Assess distance travelled during 6-minute walk tests performed with and without device. | 6 months
  Distances travelled during two six minute walk tests will be measured. Investigator will compare distance travelled with use of the device to the distance travelled without the use of the device.

SECONDARY OUTCOMES:
Assess for patient improvement in shortness of breath scores | 6 months
  This will be be measured via survey tool Borg Scale of Dyspnea (0 - no dyspnea, through 10 - maximal dyspnea). Patient scores will be measured during exercise testing with and without the device. Improvement will be considered a lower score on the Borg Scale.

CONTACTS AND LOCATIONS:
Overall Officials: John Hansen-Flaschen, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- John Hansen-Flaschen, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No